CLINICAL TRIAL: NCT03479333
Title: Short vs Standard Implants in Maxilla: a Randomized Clinical Trial
Brief Title: Short vs Standard Implants in Maxilla
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Maximiliano Sergio Cenci, Professor, Federal University of Pelotas
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PPGO025
Record Dates: First submitted 2018-03-21; First posted 2018-03-27 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Dental Implant

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short implant (Experimental)
  Interventions: Device: Short implant
- standard implant with sinus lift (Active Comparator)
  Interventions: Device: Standard implant with sinus lift

INTERVENTIONS:
Device: Short implant — Short implant will be placed depending on the previous randomization. For that, a surgical access will be done, and the implant will be placed, cover screw will be installed and the access closed. The patient will receive the definitive crown after five months after the short implant installation.
  Arms: Short implant
Device: Standard implant with sinus lift — First, a surgical access will be performed, followed by sinus lift procedure. Next, a standard implant will be placed, cover screw will be installed and the access closed. The patient will receive the definitive crown after five months after the short implant installation.
  Arms: standard implant with sinus lift

SUMMARY:
The prosthetic treatment with dental implants is challenging in posterior maxilla, where there is a sinus pneumatization. For the rehabilitation of patients with intermediate bone level, short implants have been used as alternative. It is also needed to look for the prosthetic context of rehabilitation with implants, like the use of different materials as abutments. The aim of this study is to compare the survival of two sizes of implants (short vs standard) placed in upper premolars region with need of bone graft, with a minimum of three years of follow-up, and assess the behavior of different abutments (titanium vs zirconia) in prosthesis in this context. This will be a randomized clinical trial with two groups: 1) standard implants and sinus lift; and 2) short implants without sinus lift. The patients who fulfill the inclusion criteria and accept to participate of this study, will be included in the randomization process. At the implant installation, a brown envelope, with the word SHORT or STANDARD, will be open, in order to determine the group. Abutment type will be also randomized. Four months after the installation, torque will be confirmed and the abutment will be installed. Implant failure and prosthesis failure in function of the abutment will be the outcomes. Data analysis will be conducted following a previously established spreadsheet using the Kaplan-Meier method and log rank test for success and survival, followed by Cox regression, if possible and according to the number of failures.

ELIGIBILITY:
Inclusion Criteria:

* good general and dental health;
* minimum of 6 mm bone width (BP);
* bone height in sinus region between 5 and 9 mm;
* bilateral posterior occlusal contact.

Exclusion Criteria:

* removable or partial denture;
* patient with systemic disease treatment in course;
* pregnant women;
* recent extraction at the site to receive the implant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
implant survival | five months after the implant placement
  survival will be evaluated by osseointegration presence.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Pelotas - School of Dentistry, Pelotas, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No